CLINICAL TRIAL: NCT02033759
Title: A Study of Patient Anxiety Associated With Lymphedema Surveillance: Comparing Volumetric Analysis and Bio-Impedance Analysis
Brief Title: Patient Anxiety Associated With Lymphedema Surveillance Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Research (Other)
Responsible Party: Principal Investigator, Sarah Stolker, Physical Therapist, Mercy Integrative Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Anxiety & Lymphedema
Record Dates: First submitted 2014-01-07; First posted 2014-01-13 (Estimated); Results first posted 2020-05-27 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Anxiety
Keywords: Lymphedema
MeSH Terms: conditions — Anxiety Disorders; Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional circumferential measurements (Active Comparator): Traditional screening with volumetric analysis Patient Anxiety Questionnaire
  Interventions: Other: Anxiety Questionnaire; Other: Traditional Circumferential Measurements
- Bio-Impedance Testing (Experimental): Traditional Screening with Volumetric Analysis and Bio-Impedance Analysis Patient Anxiety Questionnaire
  Interventions: Device: Bio-Impedance Testing; Other: Anxiety Questionnaire; Other: Traditional Circumferential Measurements

INTERVENTIONS:
Device: Bio-Impedance Testing — Participants in the BIA Arm will also undergo bio-impedance testing with this device.
  Other Names: LTU-400 by Impedimed
  Arms: Bio-Impedance Testing
Other: Anxiety Questionnaire — 21 item questionnaire
  Other Names: Beck Anxiety Inventory will be administered.
Other: Traditional Circumferential Measurements

SUMMARY:
We propose to study the impact of BIA screening on anxiety and primary prevention strategies for lymphedema development among patients with recent surgery for breast cancer. Currently, professional societies recommend scheduled follow-up visits to screen for lymphedema after recovery from breast cancer (e.g., 6-week, 3-month, 6-month visits with a certified lymphedema therapist). Screening involves a discussion of lymphedema symptoms and risk reduction strategies, measurement of the affected limb with a tape measure, and physical inspection for physical changes consistent with lymphedema. In the proposed study, patients will be randomly assigned to the addition of BIA screening vs. usual care. At each screening visit, all patients will be assessed for their current lymphedema risk behaviors, as outlined by the National Lymphedema Network (7). To evaluate anxiety levels, all patients will be asked to fill out the Beck Anxiety Inventory, a validated screening tool used in prior studies of patients with breast cancer (8,9). This questionnaire will be administered at each follow-up lymphedema screening visit, and the baseline will be administered at the preoperative visit. For patients randomly assigned to BIA screening, this involves the placement of adhesive electrodes on the each wrist and an ankle, followed by connection of the electrodes to the BIA machine, which then uses a painless electrical impulse to measure impedance of flow and thus asymmetry in the extracellular lymphedema volume between the 2 upper limbs (6,10). Statistical analysis will involve comparison of lymphedema risk behaviors and anxiety levels between those patients with vs. without BIA screening.

ELIGIBILITY:
Inclusion Criteria:

* Women recently diagnosed with breast cancer Age 18 and older

Exclusion Criteria:

- Those women with a pacemaker

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-06; Primary Completion 2016-09 (Actual); Study Completion 2019-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mercy Clarkson/Clayton, Creve Coeur, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
POSTER PRESENTATION AT ACRM CONFERENCE CHICAGO NOV 2016

RESULTS

PARTICIPANT FLOW:
Groups:
- Traditional Circumferential Measurements: Traditional screening with volumetric analysis Patient Anxiety Questionnaire
  Anxiety Questionnaire: 21 item questionnaire
  Traditional Circumferential Measurements
- Bio-Impedance Testing: Traditional Screening with Volumetric Analysis and Bio-Impedance Analysis Patient Anxiety Questionnaire
  Bio-Impedance Testing: Participants in the BIA Arm will also undergo bio-impedance testing with this device.
  Anxiety Questionnaire: 21 item questionnaire
  Traditional Circumferential Measurements
Period: Overall Study
Arm/Group | Traditional Circumferential Measurements | Bio-Impedance Testing
Started | 22 | 21
Completed | 19 | 19
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Traditional Circumferential Measurements: Traditional screening with volumetric analysis Patient Anxiety Questionnaire
  Anxiety Questionnaire: 21 item questionnaire
  Traditional Circumferential Measurements
  Traditional screening involved circumferential measurements using a tape measure, every 4cm from the wrist to the axilla, after which a standardized computer algorithm calculated limb volume in milliliters. Significant changes were defined as >3% volume increase when compared with the preoperative baseline limb measurements, without other clear explanation (commonly accepted unilateral volume change according to the International Society of Lymphology).
- Bio-Impedance Testing: Traditional Screening with Volumetric Analysis and Bio-Impedance Analysis Patient Anxiety Questionnaire
  Bio-Impedance Testing: Participants in the BIA Arm will also undergo bio-impedance testing with this device.
  Anxiety Questionnaire: 21 item questionnaire
  BIS measurements involved the placement of adhesive electrodes on each wrist and the right ankle, followed by connection of the electrodes to the BIS machine (L-Dex U-400, ImpediMed Ltd). The L-Dex uses a painless electrical impulse to measure impedance of flow and thus asymmetry in the extracellular lymphedema volume between the 2 upper limbs.6, 9-13 This tool compares readings to normative data to determine if significant asymmetry exists, or if the current reading is >2 standard deviations from the baseline reading for that individual.
- Total: Total of all reporting groups
Arm/Group | Traditional Circumferential Measurements | Bio-Impedance Testing | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants] — Population: Patient was excluded due to exclusion criteria
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 13 | 11 | 24
    >=65 years | 6 | 8 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38
Body Mass Index [Mean (Full Range); unit: BMI (kg/m^2) Average] | 30 [24 to 40] | 29 [21 to 42] | 30 [21 to 42]
Anxiety [Mean (Full Range); unit: units on a scale] — The Beck Anxiety Score is a measurement on a scale from 0 to 63 obtained by using the Beck Anxiety Inventory tool to assess symptoms of anxiety. A higher score correlates to increased anxiety whereas a lower score expresses a lower amount of anxiety.
  units on a scale | 7.2 [0 to 25] | 12.2 [0 to 34] | 9.6 [0 to 34]

OUTCOME MEASURES:

1. Primary Outcome: Anxiety
Description: The Beck Anxiety Score is a measurement on a scale from 0 to 63 obtained by using the Beck Anxiety Inventory tool to assess symptoms of anxiety. A higher score correlates to increased anxiety whereas a lower score expresses a lower amount of anxiety.
Time Frame: 6 weeks post-op
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Traditional Circumferential Measurements | Bio-Impedance Testing
Number analyzed (Participants) | 19 | 19
units on a scale | 7.1 [0 to 23] | 8.8 [0 to 31]

2. Primary Outcome: Anxiety
Description: as for outcome 1
Time Frame: 3 months post-op
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Traditional Circumferential Measurements | Bio-Impedance Testing
Number analyzed (Participants) | 19 | 19
units on a scale | 7.8 [0 to 26] | 10.1 [0 to 39]

3. Primary Outcome: Anxiety
Description: as for outcome 1
Time Frame: 6 months post-op
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Traditional Circumferential Measurements | Bio-Impedance Testing
Number analyzed (Participants) | 19 | 19
units on a scale | 5.1 [0 to 15] | 6.6 [0 to 20]

ADVERSE EVENTS:
Arm/Group | Traditional Circumferential Measurements | Bio-Impedance Testing
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

LIMITATIONS AND CAVEATS:
Our study used the Beck Anxiety Inventory, with its greater focus on physical symptoms of anxiety, and this approach may not have been as sensitive for identifying emotional distress when compared with other psychological tools.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No